CLINICAL TRIAL: NCT04269499
Title: Real-time MR Imaged Treatment With Holmium Microspheres of Patients With Primary or Secondary Liver Cancer; a Feasibility Study
Brief Title: Real-time Imaging of Holmium Radioembolization: a Feasibility Study
Acronym: Emeritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Quirem Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18100 Emeritus
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Liver Cancer; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm, interventional, feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients (Other): All patients receive holmium radioembolization as per usual
  Interventions: Device: QuiremSpheres®

INTERVENTIONS:
Device: QuiremSpheres® — Radioembolization with QuiremSpheres® under MR imaging

SUMMARY:
This is a feasibility study in which patients with liver tumors are treated with holmium radioembolization under real time MR imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent.
2. Female or male aged 18 years and over.
3. Diagnosis of hepatocellular carcinoma or cholangiocarcinoma in the liver or diagnosis of metastatic malignancy to the liver (primary tumours: colorectal cancer, melanoma, breast cancer or neuro-endocrine tumour) with limited disease outside the liver (i.e. liver-dominant disease) defined as the sum of the diameters of all metastases in the liver be more than 200% of the sum of the diameters of all soft tissue lesions outside the liver.
4. Patient is not amenable for standard therapies (other than radioembolisation) or patient refuses standard therapies
5. Life expectancy of 12 weeks or longer.
6. World Health Organisation (WHO) Performance status 0-1 (see Appendix III).
7. One or more measurable lesions of at least 10 mm in the longest diameter by spiral CT according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.
8. Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

1. Brain metastases or spinal cord compression, unless irradiated at least 4 weeks prior to the date of the experimental treatment and stable without steroid treatment for at least 1 week
2. Radiation therapy within the last 4 weeks before the start of study therapy.
3. The last dose of prior systemic therapy has been received less than 4 weeks prior the start of study therapy.
4. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
5. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 4.0, see Appendix II) grade 2 from previous anti-cancer therapy.
6. Serum bilirubin > 1.5 x Upper Limit of Normal (ULN).
7. Glomerular filtration rate <35 ml/min, determined according to the Modification of Diet in Renal Disease formula.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) > 5 x ULN.
9. Leukocytes < 4.0 109/l and/or platelet count < 60 109/l.
10. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
11. Pregnancy or breast feeding (women of child-bearing potential).
12. Patients suffering from diseases with an increased chance of liver toxicity, such as primary biliary cirrhosis or xeroderma pigmentosum.
13. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
14. Patients ineligible to undergo MR imaging.
15. Patients who are claustrophobic.
16. Patient who had prior liver resection and/or coil placement inside the liver, expected to cause imaging artefacts on MRI that will limit MR quantification.
17. Patients who are declared incompetent.
18. Previous enrolment in the present study or previous treatment with radioembolisation.
19. Portal vein thrombosis (tumour and/or bland) of the main branch (diagnosed on contrast enhanced transaxial images). Involvement of the right or left portal vein branches and more distal is accepted.
20. Evidence of untreated, clinically significant grade 3 portal hypertension (i.e. large varices at oesophago-gastro-duodenoscopy). In these cases, therapy with non-selective beta blocker (propranolol) or rubber band ligation should be instituted according to accepted guidelines. In case of small varices, prophylactic propranolol is advised.
21. Untreated active hepatitis.
22. Transjugular intrahepatic portosystemic shunt (TIPS).
23. Body weight over 150 kg (because of maximum table load).
24. Severe allergy for intravenous contrast agents used

    1. Iomeron®, because of CT evaluation, pre-treatment angiography and treatment angiography.
    2. Dotarem or Primovist, depending on the agent used at the time of treatment
25. Lung shunt >30 Gy, as calculated using scout dose SPECT/CT.
26. Uncorrectable extrahepatic deposition of scout dose activity. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of MR imaged administration of holmium microspheres | 1 month after inclusion
  Feasibility is defined as successful treatment under MRI in at least 4 of 6 patients. Unsuccessful treatment is defined as having to abort the procedure for safety reasons, judged by the interventional radiologist, and having to complete the administration of microspheres under X-ray guidance as in normal practice. Possible reasons for this are uncertainty about the location of the catheter, or luxation of the catheter as a result of transport to the MRI scanner.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 months after treatment
  Patients are followed up to 3 months after treatment, during which all adverse events are recorded.
Tumor/non-tumor ratio on MR based dosimetry | 1 month after inclusion
  MR based dosimetry is performed immediately after treatment, resulting in dose maps. The dose that the tumor received is divided over the dose that the rest of the liver received.
Comparison of dosimetry in Gray between MR based and SPECT based dose maps | 1 month after inclusion
  Voxel-based dosimetry will be performed, leading to dose-volume histograms with a dose value per voxel in Gray. Statistical testing will be done for differences between these data sets, i.e. the two different imaging modalities (MR based and SPECT based). It is expected that dose-volume histograms will be similar between the two modalities.
Tumor response after 3 months based on CT imaging (according to RECIST 1.1 criteria) | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank Nijsen, PhD, Principal Investigator — Associate professor
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van den Brekel A, Snoeijink TJ, de Meijer VE, Boswinkel M, de Jong KP, Roosen J, Arranja AG, Futterer JJ, Ruiter SJS, Nijsen JFW. Spatial distribution of fractionally administered holmium microspheres in non-tumorous human liver tissue: how livers survive transarterial radioembolisation. EJNMMI Res. 2025 Apr 28;15(1):49. doi: 10.1186/s13550-025-01240-8. PMID 40289050
- [Derived] Roosen J, Westlund Gotby LEL, Arntz MJ, Futterer JJ, Janssen MJR, Konijnenberg MW, van Wijk MWM, Overduin CG, Nijsen JFW. Intraprocedural MRI-based dosimetry during transarterial radioembolization of liver tumours with holmium-166 microspheres (EMERITUS-1): a phase I trial towards adaptive, image-controlled treatment delivery. Eur J Nucl Med Mol Imaging. 2022 Nov;49(13):4705-4715. doi: 10.1007/s00259-022-05902-w. Epub 2022 Jul 13. PMID 35829749